CLINICAL TRIAL: NCT05623787
Title: Diagnostic Value of Diffusion-weighted Magnetic Resonance Imaging for Detection of Peritoneal Recurrence in Patients With High-risk Colorectal and Appendiceal Neoplasms : a Pilot Study
Brief Title: Diagnostic Value of Diffusion-weighted Magnetic Resonance in High-risk Colorectal and Appendiceal Neoplasms
Acronym: DWI-HighRisk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Alexandre Brind'Amour, Doctor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MP-20-2022-6366
Record Dates: First submitted 2022-11-10; First posted 2022-11-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Peritoneal Carcinomatosis; Peritoneal Metastases; Appendix Cancer; Appendix Neoplasm; Colorectal Cancer
Keywords: DWI; CRC; Carcinomatosis; Diagnostic laparoscopy
MeSH Terms: conditions — Peritoneal Neoplasms; Appendiceal Neoplasms; Colorectal Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DWI-High Risk (Experimental): Patients to undergo DWI-MRI (patients included in the study).
  Interventions: Diagnostic Test: Whole-body diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Whole-body diffusion-weighted magnetic resonance imaging — See arm description.

SUMMARY:
Diffusion-weighted magnetic resonance imaging (DWI/MRI) has been described in recent literature as a highly sensitive and specific modality for the detection of peritoneal metastases PM. It has been demonstrated to be superior to CT for patients with known peritoneal disease from colorectal and gynaecological malignancies as a staging tool for cytoreductive surgery. It was also demonstrated to be superior for the detection of PM for gastric cancer patients otherwise considered with a resectable tumor. However, the literature is scarce on the role of DWI/MRI in the detection of peritoneal recurrence for patients with high-risk features, either colorectal cancer (CRC) or appendiceal neoplasms (AN).

The aim of this study is to prospectively assess the added value of whole-body DWI/MRI (WB-DWI/MRI) to CT and diagnostic laparoscopy for detection of PM in the follow-up of patients presenting with CRC or AN and high-risk features for peritoneal recurrence and evaluate how it correlates with intraoperative findings.

DETAILED DESCRIPTION:
This is a multicentric, prospective study (CHU de Québec and Hôpital Maisonneuve-Rosemont). Patients will be referred to one of six surgeons with a subspeciality in peritoneal surface oncology after their index surgery for CRC or AN. After thorough assessment, patients judged without residual peritoneal disease, but at high-risk for peritoneal recurrence, will be prospectively included in the study. Patients will be assessed with CT and WB-DWI/MRI twelve months after their index surgery. For WB-DWI/MRI, the standard protocol will include the following sequences: Patients will drink 1L of pineapple juice one hour prior to the examination in order to provide a negative intraluminal contrast. They will receive 20 mg of intravenous hyoscine butylbromide at the beginning of the MR exam in order to reduce bowel peristalsis. Sequences will include Axial et Coronal T2WI of the abdomen and pelvis, axial DWI with b values of 0, 50 and 1000 of the abdomen and pelvis, as well as Pre and post gadolinium-based contrast Axial and Coronal 3D T1WGRE. All patients included in the study will then undergo diagnostic laparoscopy, to provide correlation with imaging findings. Patients with no evidence of peritoneal recurrence on CT, WB-DWI/MRI and diagnostic laparoscopy will continue to be followed with serial CT and blood tumor markers (CEA, CA 19-9) as done on a routine basis. Patients with confirmed peritoneal disease at diagnostic laparoscopy will be further evaluated for cytoreductive surgery, with or without hyperthermic intraperitoneal chemotherapy. The study duration will be two years for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of colorectal cancer or high-risk appendiceal neoplasm (High grade Appendiceal Mucinous Neoplasm (HAMN), goblet-cell carcinoma or adenocarcinoma).
* No evidence of residual peritoneal disease based on referring surgeon operating report and preoperative imaging.
* At least one high-risk feature for peritoneal recurrence, including:

  * Synchronous peritoneal metastases resected at index surgery;
  * Synchronous ovarian metastases resected at index surgery;
  * Perforated primary tumor.
* No evidence of distant metastases.
* Patient fit for cytoreductive surgery, if required (ECOG 0 or 1).

Exclusion Criteria:

* Unresected synchronous peritoneal metastases at referral.
* Low grade Appendiceal Mucinous Neoplasm (LAMN).
* No high-risk feature for peritoneal recurrence.
* Evidence of distant metastases on preoperative imaging.
* Patient who is unable to have MRI.
* Patient unfit for cytoreductive surgery, if required (ECOG 2 or more).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Peritoneal findings | 24 months
  The number of cases in which peritoneal findings on MRI matched with surgical exploration.
Early peritoneal recurrence | 36 months
  The number of cases with early peritoneal recurrence after MRI.

SECONDARY OUTCOMES:
Early distant recurrence | 36 months
  The number of cases with early distant recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Brind'Amour, MD, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - CHU de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Massalou D, Benizri E, Chevallier A, Duranton-Tanneur V, Pedeutour F, Benchimol D, Bereder JM. Peritoneal carcinomatosis of colorectal cancer: novel clinical and molecular outcomes. Am J Surg. 2017 Feb;213(2):377-387. doi: 10.1016/j.amjsurg.2016.03.008. Epub 2016 Aug 5. PMID 27816197
- [Background] Sugarbaker PH. Colorectal cancer: prevention and management of metastatic disease. Biomed Res Int. 2014;2014:782890. doi: 10.1155/2014/782890. Epub 2014 Mar 24. PMID 24783222
- [Background] Goere D, Glehen O, Quenet F, Guilloit JM, Bereder JM, Lorimier G, Thibaudeau E, Ghouti L, Pinto A, Tuech JJ, Kianmanesh R, Carretier M, Marchal F, Arvieux C, Brigand C, Meeus P, Rat P, Durand-Fontanier S, Mariani P, Lakkis Z, Loi V, Pirro N, Sabbagh C, Texier M, Elias D; BIG-RENAPE group. Second-look surgery plus hyperthermic intraperitoneal chemotherapy versus surveillance in patients at high risk of developing colorectal peritoneal metastases (PROPHYLOCHIP-PRODIGE 15): a randomised, phase 3 study. Lancet Oncol. 2020 Sep;21(9):1147-1154. doi: 10.1016/S1470-2045(20)30322-3. Epub 2020 Jul 24. PMID 32717180
- [Background] Klaver CEL, Wisselink DD, Punt CJA, Snaebjornsson P, Crezee J, Aalbers AGJ, Brandt A, Bremers AJA, Burger JWA, Fabry HFJ, Ferenschild F, Festen S, van Grevenstein WMU, Hemmer PHJ, de Hingh IHJT, Kok NFM, Musters GD, Schoonderwoerd L, Tuynman JB, van de Ven AWH, van Westreenen HL, Wiezer MJ, Zimmerman DDE, van Zweeden AA, Dijkgraaf MGW, Tanis PJ; COLOPEC collaborators group. Adjuvant hyperthermic intraperitoneal chemotherapy in patients with locally advanced colon cancer (COLOPEC): a multicentre, open-label, randomised trial. Lancet Gastroenterol Hepatol. 2019 Oct;4(10):761-770. doi: 10.1016/S2468-1253(19)30239-0. Epub 2019 Jul 29. PMID 31371228
- [Background] Honore C, Goere D, Souadka A, Dumont F, Elias D. Definition of patients presenting a high risk of developing peritoneal carcinomatosis after curative surgery for colorectal cancer: a systematic review. Ann Surg Oncol. 2013 Jan;20(1):183-92. doi: 10.1245/s10434-012-2473-5. Epub 2012 Oct 23. PMID 23090572
- [Background] Soucisse ML, Lansom J, Alshahrani MS, Morris DL. Mucinous appendiceal neoplasms with or without pseudomyxoma peritonei: a review. ANZ J Surg. 2020 Oct;90(10):1888-1894. doi: 10.1111/ans.16185. Epub 2020 Aug 5. PMID 32761790
- [Background] Chicago Consensus Working Group. The Chicago Consensus on Peritoneal Surface Malignancies: Management of Appendiceal Neoplasms. Ann Surg Oncol. 2020 Jun;27(6):1753-1760. doi: 10.1245/s10434-020-08316-w. Epub 2020 Apr 13. PMID 32285275
- [Background] Chua TC, Moran BJ, Sugarbaker PH, Levine EA, Glehen O, Gilly FN, Baratti D, Deraco M, Elias D, Sardi A, Liauw W, Yan TD, Barrios P, Gomez Portilla A, de Hingh IH, Ceelen WP, Pelz JO, Piso P, Gonzalez-Moreno S, Van Der Speeten K, Morris DL. Early- and long-term outcome data of patients with pseudomyxoma peritonei from appendiceal origin treated by a strategy of cytoreductive surgery and hyperthermic intraperitoneal chemotherapy. J Clin Oncol. 2012 Jul 10;30(20):2449-56. doi: 10.1200/JCO.2011.39.7166. Epub 2012 May 21. PMID 22614976
- [Background] Tiselius C, Kindler C, Shetye J, Letocha H, Smedh K. Computed Tomography Follow-Up Assessment of Patients with Low-Grade Appendiceal Mucinous Neoplasms: Evaluation of Risk for Pseudomyxoma Peritonei. Ann Surg Oncol. 2017 Jul;24(7):1778-1782. doi: 10.1245/s10434-016-5623-3. Epub 2017 May 4. PMID 28474197
- [Background] Hegg KS, Mack LA, Bouchard-Fortier A, Temple WJ, Gui X. Macroscopic and microscopic characteristics of low grade appendiceal mucinous neoplasms (LAMN) on appendectomy specimens and correlations with pseudomyxoma peritonei development risk. Ann Diagn Pathol. 2020 Oct;48:151606. doi: 10.1016/j.anndiagpath.2020.151606. Epub 2020 Aug 21. PMID 32889392
- [Background] Reiter S, Rog CJ, Alassas M, Ong E. Progression to pseudomyxoma peritonei in patients with low grade appendiceal mucinous neoplasms discovered at time of appendectomy. Am J Surg. 2022 Jun;223(6):1183-1186. doi: 10.1016/j.amjsurg.2021.12.003. Epub 2021 Dec 3. PMID 34879923
- [Background] Orr CE, Yantiss RK. Controversies in appendiceal pathology: mucinous and goblet cell neoplasms. Pathology. 2022 Mar;54(2):167-176. doi: 10.1016/j.pathol.2021.09.003. Epub 2021 Nov 23. PMID 34836648
- [Background] Elekonawo FMK, Starremans B, Laurens ST, Bremers AJA, de Wilt JHW, Heijmen L, de Geus-Oei LF. Can [18F]F-FDG PET/CT be used to assess the pre-operative extent of peritoneal carcinomatosis in patients with colorectal cancer? Abdom Radiol (NY). 2020 Feb;45(2):301-306. doi: 10.1007/s00261-019-02268-w. PMID 31642963
- [Background] Esquivel J, Chua TC, Stojadinovic A, Melero JT, Levine EA, Gutman M, Howard R, Piso P, Nissan A, Gomez-Portilla A, Gonzalez-Bayon L, Gonzalez-Moreno S, Shen P, Stewart JH, Sugarbaker PH, Barone RM, Hoefer R, Morris DL, Sardi A, Sticca RP. Accuracy and clinical relevance of computed tomography scan interpretation of peritoneal cancer index in colorectal cancer peritoneal carcinomatosis: a multi-institutional study. J Surg Oncol. 2010 Nov 1;102(6):565-70. doi: 10.1002/jso.21601. PMID 20976729
- [Background] Elias D, Honore C, Dumont F, Ducreux M, Boige V, Malka D, Burtin P, Dromain C, Goere D. Results of systematic second-look surgery plus HIPEC in asymptomatic patients presenting a high risk of developing colorectal peritoneal carcinomatosis. Ann Surg. 2011 Aug;254(2):289-93. doi: 10.1097/SLA.0b013e31822638f6. PMID 21709543
- [Background] Elias D, Gilly F, Boutitie F, Quenet F, Bereder JM, Mansvelt B, Lorimier G, Dube P, Glehen O. Peritoneal colorectal carcinomatosis treated with surgery and perioperative intraperitoneal chemotherapy: retrospective analysis of 523 patients from a multicentric French study. J Clin Oncol. 2010 Jan 1;28(1):63-8. doi: 10.1200/JCO.2009.23.9285. Epub 2009 Nov 16. PMID 19917863
- [Background] Chua TC, Morris DL, Esquivel J. Impact of the peritoneal surface disease severity score on survival in patients with colorectal cancer peritoneal carcinomatosis undergoing complete cytoreduction and hyperthermic intraperitoneal chemotherapy. Ann Surg Oncol. 2010 May;17(5):1330-6. doi: 10.1245/s10434-009-0866-x. Epub 2009 Dec 22. PMID 20033321
- [Background] Brind'Amour A, Dube P, Tremblay JF, Soucisse ML, Mack L, Bouchard-Fortier A, McCart JA, Govindarajan A, Bischof D, Haase E, Giacomantonio C, Hebbard P, Younan R, MacNeill A, Boulanger-Gobeil C, Sideris L. Canadian guidelines on the management of colorectal peritoneal metastases. Curr Oncol. 2020 Dec;27(6):e621-e631. doi: 10.3747/co.27.6919. Epub 2020 Dec 1. PMID 33380878
- [Background] Dong L, Li K, Peng T. Diagnostic value of diffusion-weighted imaging/magnetic resonance imaging for peritoneal metastasis from malignant tumor: A systematic review and meta-analysis. Medicine (Baltimore). 2021 Feb 5;100(5):e24251. doi: 10.1097/MD.0000000000024251. PMID 33592867
- [Background] Dresen RC, De Vuysere S, De Keyzer F, Van Cutsem E, Prenen H, Vanslembrouck R, De Hertogh G, Wolthuis A, D'Hoore A, Vandecaveye V. Whole-body diffusion-weighted MRI for operability assessment in patients with colorectal cancer and peritoneal metastases. Cancer Imaging. 2019 Jan 7;19(1):1. doi: 10.1186/s40644-018-0187-z. PMID 30616608
- [Background] Zhang H, Dai W, Fu C, Yan X, Stemmer A, Tong T, Cai G. Diagnostic value of whole-body MRI with diffusion-weighted sequence for detection of peritoneal metastases in colorectal malignancy. Cancer Biol Med. 2018 May;15(2):165-170. doi: 10.20892/j.issn.2095-3941.2017.0162. PMID 29951340
- [Background] Namimoto T, Awai K, Nakaura T, Yanaga Y, Hirai T, Yamashita Y. Role of diffusion-weighted imaging in the diagnosis of gynecological diseases. Eur Radiol. 2009 Mar;19(3):745-60. doi: 10.1007/s00330-008-1185-5. Epub 2008 Oct 7. PMID 18839179
- [Background] van 't Sant I, van Eden WJ, Engbersen MP, Kok NFM, Woensdregt K, Lambregts DMJ, Shanmuganathan S, Beets-Tan RGH, Aalbers AGJ, Lahaye MJ. Diffusion-weighted MRI assessment of the peritoneal cancer index before cytoreductive surgery. Br J Surg. 2019 Mar;106(4):491-498. doi: 10.1002/bjs.10989. Epub 2018 Oct 24. PMID 30353920
- [Background] De Vuysere S, Vandecaveye V, De Bruecker Y, Carton S, Vermeiren K, Tollens T, De Keyzer F, Dresen RC. Accuracy of whole-body diffusion-weighted MRI (WB-DWI/MRI) in diagnosis, staging and follow-up of gastric cancer, in comparison to CT: a pilot study. BMC Med Imaging. 2021 Feb 5;21(1):18. doi: 10.1186/s12880-021-00550-2. PMID 33546626